CLINICAL TRIAL: NCT04119791
Title: A Multidisciplinary Investigation of Cardiovascular Benefits of Wild Rice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Mohammed Moghadasian, Principal Investigator, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS22890
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Healthy Diet; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wild rice (Experimental): Participants will consume one serving of the test food containing wild rice every day over 28 days.
  Interventions: Other: wild rice

INTERVENTIONS:
Other: wild rice — 30 grams of wild rice in the form salad, snack bar and soup

SUMMARY:
In this study 24 adult males and adult females, with overall healthy condition, will consume approximately 30 grams of wild rice every day for 28 days. Cardiovascular risk factors will be assessed at the beginning and at the end of the study.

DETAILED DESCRIPTION:
Cardiovascular disorders (CVD) including hypertension, myocardial infarction and stroke are still among the top causes of mortality and morbidity in both developed and developing countries. Several modifiable and non-modifiable risk factors play a crucial role in pathogenesis of CVD. Among modifiable risk factors, unhealthy diets and sedentary life style have been recognized worldwide. In this regard, many health authorities have developed guidelines to promote consumption of healthy diets and an active life style among the general population and for CVD patients. Furthermore, recent advances in the area of food and nutrition have revealed health promoting properties for some foods beyond their nutritional values. Such foods are generally known as "functional foods." The Department of Food and Human Nutritional Sciences at the University of Manitoba (U of M) is well-recognized for its contribution in this area of research. However, the effects of wild rice have not been tested in clinical trials. Hence, a pilot study is required before performing a large clinical trial to explore the effects of wild rice consumption and its potential mechanisms. This would not only benefit the populations, but also warranty its scope globally. In this study, the investigators will carry out such a study on the cardiovascular benefits of wild rice in 24 women and 24 men (20-40 years old) over a period of 4 weeks. "Test food" including fruit/vegetable salad, energy cookies and casserole will be prepared by Tall Grass Bakery, Winnipeg, Manitoba. These foods will contain approximately 30 grams of wild rice per serving. The participants will be recruited per our standard procedures. After completion of recruitment procedures, including obtaining a fully informed consent form and health information, the participant will be asked to consume one serving of the "test food" every day over 28 days. Vascular measurements, plus urine and blood samples will be collected at day 0 and day 28. Serum lipids, inflammatory markers and fecal bacterial type, and numbers will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Female
* Both genders are healthy
* 20 - 40 years old

Exclusion Criteria:

* Non-pregnant
* Non-lactating
* Non-smokers
* Not obese (Body Mass Index (BMI) < 30)
* Not currently on any medications for cardiovascular, diabetes, and cancer diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult 20 - 40 years of age
Enrollment: 48 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Wild rice alters gut microbiome. | 4 weeks
  This study is designed to investigate the effects of wild rice consumption on gut microbiome diversity and population in volunteer healthy young adults.
Changes in gut microbiome alters macronutrient metabolism. | 4 weeks
  In this study, the investigators will establish whether changes in gut microbiome due to consumption of wild rice may result in altered macronutrient metabolism by studying plasma metabolomics.

SECONDARY OUTCOMES:
Wild rice consumption improves blood lipid profile. | 4 weeks
  In this study, plasma lipoprotein cholesterol concentrations will be estimated to assess the impact of wild rice consumption on the overall risk for atherosclerosis.
Will rice consumption improves endothelial cell function. | 4 weeks
  Mobil-O-Graph techniques will be used to measure endothelial cell function in the participants prior to consumption of wild rice and after 28 days of consumption of wild rice. This study will establish the effects of wild rice consumption on endothelial cell function.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed H Moghadasian, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital Research Center Asper clinical, Winnipeg, Manitoba, Canada